CLINICAL TRIAL: NCT04605042
Title: A Multicenter Prospective Clinical Study of Wet-suction Technique and Standard Negative Pressure Technique in EUS-FNB for the Diagnosis of Pancreatic Solid Mass
Brief Title: Comparsion of WT and SNP Techniques of EUS-FNB in Pancreatic Solid Mass (WESP-PSM)
Acronym: WESP-PSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Changhai Hospital (Other); Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, duowu zou, prof. and director, Ruijin Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: RuijinH2020301
Record Dates: First submitted 2020-10-01; First posted 2020-10-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Pancreatic Neoplasms; Diagnoses Disease
Keywords: endoscopic ultrasound; endoscopic ultrasound guided FNB
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WET First group (Experimental): COOK ECHO-HD 22-C EchoTip Procore needle biopsy in WS-SNP-WS-SNP sequence
  Interventions: Procedure: wet suction; Procedure: standard negative pressure suction
- STANDARD first group (Experimental): COOK ECHO-HD 22-C EchoTip Procore needle in SNP-WS-SNP-WS sequence
  Interventions: Procedure: wet suction; Procedure: standard negative pressure suction

INTERVENTIONS:
Procedure: wet suction — Before pucturing the lesion, the stylet was removed and the needle was pre-flushed with 1-2 mL of saline using a 10-mL syringe, the endoscopist then punctured the lesion and replaced the 10-mL syringe with a 10-mL pre-vacuum syringe
Procedure: standard negative pressure suction — after puncturing the lesion, the endoscopist removed the stylet and attached a 10-mL pre-vacuum syringe for aspiration.

SUMMARY:
The purpose of this study is to compare the diagnosis accuracy between of wet suction (WS) technique and standard negative pressure (SNP) technique in EUS-FNB by 22G EUS Procore fine needle biopsy（FNB）device for solid pancreatic lesions.

DETAILED DESCRIPTION:
This is a multi-center, single-blind, randomized, controlled trial. two hundred and ninety six patients with solid pancreatic lesions referred for EUS guided fine needle biopsy will be randomly assigned to two groups. For group A which will be used with 22G EUS Procore fine needle biopsy device, the pass sequence is WS-SNP-WS-SNP technique. For group B with 22G EUS Procore fine needle biopsy device, the pass sequence is SNP-WS-SNP-WS. All procedures will be performed by experienced echo-endoscopists, and the patients and assessors (cytologists and pathologists) will be blinded during the entire study. The primary outcome measure is the diagnosis yield. Secondary outcome measures are specimen quality.

ELIGIBILITY:
Inclusion Criteria:

1. informed consent
2. Subjects over 18 years old
3. Imaging examination (ultrasound, CT or MRI) diagnosed or suspected solid pancreatic mass more than 1cm

Exclusion Criteria:

1. Unable or refused to sign informed consent
2. suspended anticoagulant/antiplatelet therapy
3. Being pregnant or breastfeeding
4. Cystic lesions of the pancreas
5. coagulation disorders (PLT <50×103/ L, INR > 1.5)
6. A history of mental illness
7. other medical conditions that are not suitable for FNB puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic sensitivity of WS technique and SNP technique by EUS-FNB | 6 month
  Sensitivity will be calculated as the probability of actually having pancreatic diasease and being diagnosed by WS technique during EUS-FNB
diagnostic specificity of WS technique and SNP technique by EUS-FNB | 6 month
  specificity will be calculated as the probability of actually not having the pancreatic disease and being diagnosed as being free of the disease by WS or SNP technique during EUS-FNB

SECONDARY OUTCOMES:
Sample adequacy of WS technique and SNP technique by EUS-FNB | 6 month
  The tissue integrity assessments of specimens will be evaluated by score 0-3. Score 3, sufficient material for adequate histological interpretation; Score 2, samples allowing limited histological assessment; Score 1,samples not providing histological information.
Cell density of WS technique and SNP technique by EUS-FNB | 6 month
  The Cell density assessments of specimens will be evaluated by score A-C. Score A：Satisfactory, more than 4 clusters of cells, each cluster more than 10 cells.
  Score B：Sufficient, approximately 2-4 clusters, each with more than 10 cells Score C: ：Unsatisfactory, less than 2 clusters or no cells on slide

CONTACTS AND LOCATIONS:
Overall Officials: DuoWu Zou, Ph.D,M.D, Study Chair — Ruijin hospital Shanghai Jiaotong Universtity, school of medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dumonceau JM, Deprez PH, Jenssen C, Iglesias-Garcia J, Larghi A, Vanbiervliet G, Aithal GP, Arcidiacono PG, Bastos P, Carrara S, Czako L, Fernandez-Esparrach G, Fockens P, Gines A, Havre RF, Hassan C, Vilmann P, van Hooft JE, Polkowski M. Indications, results, and clinical impact of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline - Updated January 2017. Endoscopy. 2017 Jul;49(7):695-714. doi: 10.1055/s-0043-109021. Epub 2017 May 16. PMID 28511234
- [Background] Banafea O, Mghanga FP, Zhao J, Zhao R, Zhu L. Endoscopic ultrasonography with fine-needle aspiration for histological diagnosis of solid pancreatic masses: a meta-analysis of diagnostic accuracy studies. BMC Gastroenterol. 2016 Aug 31;16(1):108. doi: 10.1186/s12876-016-0519-z. PMID 27580856
- [Background] Puli SR, Bechtold ML, Buxbaum JL, Eloubeidi MA. How good is endoscopic ultrasound-guided fine-needle aspiration in diagnosing the correct etiology for a solid pancreatic mass?: A meta-analysis and systematic review. Pancreas. 2013 Jan;42(1):20-6. doi: 10.1097/MPA.0b013e3182546e79. PMID 23254913
- [Background] Lee JK, Choi JH, Lee KH, Kim KM, Shin JU, Lee JK, Lee KT, Jang KT. A prospective, comparative trial to optimize sampling techniques in EUS-guided FNA of solid pancreatic masses. Gastrointest Endosc. 2013 May;77(5):745-51. doi: 10.1016/j.gie.2012.12.009. Epub 2013 Feb 21. PMID 23433878
- [Background] Moller K, Papanikolaou IS, Toermer T, Delicha EM, Sarbia M, Schenck U, Koch M, Al-Abadi H, Meining A, Schmidt H, Schulz HJ, Wiedenmann B, Rosch T. EUS-guided FNA of solid pancreatic masses: high yield of 2 passes with combined histologic-cytologic analysis. Gastrointest Endosc. 2009 Jul;70(1):60-9. doi: 10.1016/j.gie.2008.10.008. Epub 2009 Apr 25. PMID 19394012
- [Background] Sakamoto H, Kitano M, Komaki T, Noda K, Chikugo T, Dote K, Takeyama Y, Das K, Yamao K, Kudo M. Prospective comparative study of the EUS guided 25-gauge FNA needle with the 19-gauge Trucut needle and 22-gauge FNA needle in patients with solid pancreatic masses. J Gastroenterol Hepatol. 2009 Mar;24(3):384-90. doi: 10.1111/j.1440-1746.2008.05636.x. Epub 2008 Nov 20. PMID 19032453
- [Background] Polkowski M, Jenssen C, Kaye P, Carrara S, Deprez P, Gines A, Fernandez-Esparrach G, Eisendrath P, Aithal GP, Arcidiacono P, Barthet M, Bastos P, Fornelli A, Napoleon B, Iglesias-Garcia J, Seicean A, Larghi A, Hassan C, van Hooft JE, Dumonceau JM. Technical aspects of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Technical Guideline - March 2017. Endoscopy. 2017 Oct;49(10):989-1006. doi: 10.1055/s-0043-119219. Epub 2017 Sep 12. PMID 28898917
- [Background] Alatawi A, Beuvon F, Grabar S, Leblanc S, Chaussade S, Terris B, Barret M, Prat F. Comparison of 22G reverse-beveled versus standard needle for endoscopic ultrasound-guided sampling of solid pancreatic lesions. United European Gastroenterol J. 2015 Aug;3(4):343-52. doi: 10.1177/2050640615577533. PMID 26279842
- [Background] Attam R, Arain MA, Bloechl SJ, Trikudanathan G, Munigala S, Bakman Y, Singh M, Wallace T, Henderson JB, Catalano MF, Guda NM. "Wet suction technique (WEST)": a novel way to enhance the quality of EUS-FNA aspirate. Results of a prospective, single-blind, randomized, controlled trial using a 22-gauge needle for EUS-FNA of solid lesions. Gastrointest Endosc. 2015;81(6):1401-7. doi: 10.1016/j.gie.2014.11.023. Epub 2015 Feb 27. PMID 25733127
- [Background] Wang Y, Wang RH, Ding Z, Tan SY, Chen Q, Duan YQ, Zhu LR, Cao JW, Wang J, Shi G, Wu XL, Wang JL, Zhao YC, Tang SJ, Cheng B. Wet- versus dry-suction techniques for endoscopic ultrasound-guided fine-needle aspiration of solid lesions: a multicenter randomized controlled trial. Endoscopy. 2020 Nov;52(11):995-1003. doi: 10.1055/a-1167-2214. Epub 2020 May 15. PMID 32413915
- [Background] Li DF, Wang JY, Yang MF, Xiong F, Zhang DG, Xu ZL, Luo MH, Jing ZD, Wang KX, Wang LS, Yao J. Factors associated with diagnostic accuracy, technical success and adverse events of endoscopic ultrasound-guided fine-needle biopsy: A systematic review and meta-analysis. J Gastroenterol Hepatol. 2020 Aug;35(8):1264-1276. doi: 10.1111/jgh.14999. Epub 2020 Feb 23. PMID 32003100